CLINICAL TRIAL: NCT02795078
Title: To Investigate the Coexistence of Atherosclerotic Intracranial Arterial Stenosis With Intracranial Aneurysms
Brief Title: The Coexistence of Atherosclerotic Intracranial Arterial Stenosis With Intracranial Aneurysms
Acronym: CAIASA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: liuxingju (Other Government)
Collaborators: National Clinical Research Center for Neurological Diseases (Unknown)
Responsible Party: Sponsor-Investigator, liuxingju, Ministry of Science and Technology of the People´s Republic of China, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Other Study IDs: BJTTH-001
Record Dates: First submitted 2016-06-05; First posted 2016-06-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Atherosclerotic Intracranial Arterial Stenosis With Intracranial Aneurysms
Keywords: Atherosclerotic Intracranial Arterial Stenosis; Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Conservative Treatment; Stents; Constriction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: conservative treatment
Procedure: Aneurysms clipping
Procedure: Interventional embolization forAneurysms
Procedure: stenting for stenosis

SUMMARY:
Atherosclerotic intracranial arterial（ICA） stenosis and intracranial aneurysms are the common causes of ischemic stroke and hemorrhagic stroke, respectively. Investigators aimed to assess the prevalence of cerebral aneurysms in patients with atherosclerotic intracranial arterial stenosis.

DETAILED DESCRIPTION:
Based on prospective data of patients with symptomatic or asymptomatic ICA stenosis admitted to Beijing Tiantan Hospital between Jan 2015 and July 2016, all patients underwent brain CTA / MRA/DSA. Investigators determined the number of the patients with intracranial aneurysms, calculated overall prevalence of the coexistence of atherosclerotic ICA stenosis with aneurysms and analyzed the clinical features.

ELIGIBILITY:
Inclusion Criteria:

1. DSA identified the coexistence of intracranial Arterial Stenosis With Intracranial Aneurysms
2. Stenosis caused by atherosclerosis

Exclusion Criteria:

1. patients do not agree
2. Stenosis caused by no atherosclerosis disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who had the coexistence of intracranial Arterial Stenosis With Intracranial Aneurysms were included in this study
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
new stroke events during perioperative period | perioperative period

SECONDARY OUTCOMES:
stroke events during follow up | 6 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yin Z, Zhang Q, Zhao Y, Lu J, Ge P, Xie H, Wu D, Yu S, Kang S, Zhang Q, Zhang Y, Zhang D, Zhao J, Liu X. Prevalence and Procedural Risk of Intracranial Atherosclerotic Stenosis Coexisting With Unruptured Intracranial Aneurysm. Stroke. 2023 Jun;54(6):1484-1493. doi: 10.1161/STROKEAHA.122.041553. Epub 2023 May 4. PMID 37139814